CLINICAL TRIAL: NCT06723730
Title: ADDITIONAL EFFECTS OF MOBILIZATION WITH MOVEMENT WITH UPPER QUADRANT CORE STRENGTHENING IN ROTATOR CUFF RELATED PAIN:A RANDOMIZED CONTROLLED TRAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/57
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Syndrome
MeSH Terms: interventions — Movement

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Quadrant Strenghtening + MWM Group (Experimental): In addition to upper quadrant core strengthening protocol participants will also perform mobilization with movement.
  Mobilization with movement protocol will comprise of following forms.
  1. Acromioclavicular joint glides
  2. Scapular glides
  3. Glenohumeral joint glides ( inferior glides, postero-lateral glides, postero-inferior)
  Interventions: Procedure: Upper Quadrant Core Strengthening protocol; Procedure: Mobilization with movement
- Upper Quadrant Strenghtening Group (Experimental): Participants will perform upper quadrant core strengthening protocol. Upper quadrant core strengthening protocol will comprise of following four week protocol.
  1. Week One Scapular postural correction , Shoulder Shrugging exercises
  2. Week Two External rotation at 0 degree
  3. Week Three Internal rotation at 0 degree
  4. Week Four Standing Row at 45 and 90 degree, Anterior shoulder stretch , Thoracic exercises in sitting
  Interventions: Procedure: Upper Quadrant Core Strengthening protocol

INTERVENTIONS:
Procedure: Upper Quadrant Core Strengthening protocol — Upper Quadrant Core Strengthening protocol Core strengthening protocol will comprise of following four week protocol.
  1. Week one Scapular postural correction and shoulder shrugging exercises
  2. Week two External rotation at 0 degree
  3. Week three Internal rotation at 0 degree
  4. Week four Standing row at 45 and 90 degree , Anterior shoulder stretch and Thoracic exercise in sitting
Procedure: Mobilization with movement — In addition to upper quadrant core strengthening protocol participants will also perform mobilization with movement.
  Mobilization with movement protocol will comprise of following forms.
  1. Acromioclavicular joint glides
  2. Scapular glides
  3. Glenohumeral joint glides ( inferior glides, postero-lateral glides, postero-inferior)
  Arms: Upper Quadrant Strenghtening + MWM Group

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the additional effects of mobilization with movement with upper quadrant core strengthening in rotator cuff related pain

.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of mobilization with movement with upper quadrant core strengthening in rotator cuff related shoulder pain on A. Pain B. Range of motion C. Propioception D. Kinesiophobia

Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Recruited participants will be allocated to either of the groups through a sealed opaque envelope method.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Both genders
* Unilateral shoulder pain of traumatic origin
* Scoring should be less than 8 on numeric pain rating scale
* Symptoms lasting more than 6 weeks
* Pain on active shoulder movement
* Pain provoked by atleast three of the following tests. A. Neer test B. Hawkins-Kennedy test C. Empty Can test D. Full Can test E. Painfull Arc test F. Resisted external rotation test
* Patients reffered by a rehabilitation and orthopedic specialistwith diagnosis of rotator cuff injury, subacromial impingement syndrome, subacromial pain

Exclusion Criteria:

* History and Clinical presentation compatible with complete rotator cuff or bicep brachia rupture
* Adhesive capsulitis
* History of dislocation
* Glenohumeral osteoarthritis
* Cancer
* Auto-immune inflammatory conditions and infection
* Positive joint integrity tests ( Ant. and Post. Drawer tests)
* Hill sachs lesions
* Bankarts lesions
* Cervical rib
* Previous shoulder or neck surgery or fracture
* Familiar pain provoked by neck movements
* Presence of radicular sign
* Diagnosis of fibromyalgia
* Clinical depression
* Rheumatoid arthritis
* Poor bone quality ( osteoporosis)
* Vertobrobasilar insufficiency test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Pain will be measured on Numerical Pain rating scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Range of motion | 4 weeks
  A universal goniometer will be used to measure the shoulder ROM in external & internal rotation, abduction and flexion and their normal ranges are 90, 80, 0-180, 0-180 degree respectively.
Proprioception | 4 weeks
  The laser pointer method for assessing Shoulder Joint Position Sense (JPS) involves the patient using a laser pointer to target a 1 meter distanced scoreboard while performing arm movements. Patient will be asked to perform flexion, abduction and external rotation to 90 degree or alternatively to maximum possible pain free range below 90 degree. After three practice rounds with eyes open, four attempt with eye closed will be performed and shoulder range will be measured. We will measure JPSE for flexion, abduction and external rotation by using mobile app inclinometer.
Kinesiophobia | 4 Weeks
  The Tampa Scale of Kinesiophobia (TSK) is a 17-item self-report tool with a 4-point Likert scale, measuring fear of movement due to injury or pain, and somatic focus on underlying medical issues. Scores range from 17 to 68, with higher scores (≥37) indicating significant kinesiophobia and poorer health outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan